CLINICAL TRIAL: NCT03033823
Title: Multicenter Randomized Placebo Controlled Trial Assessing the Efficacy of Oral Adjuvant Magnesium Supplementation in the Treatment of Alcohol Withdrawal Syndrome
Brief Title: MAGnesium Adjunction in Alcohol Withdrawal Syndrome: a Multicenter Assessment (MAGMA)
Acronym: MAGMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150939; 2016-002072-26 (EudraCT Number); PHRC (Other Grant/Funding Number: 15-613)
Record Dates: First submitted 2017-01-03; First posted 2017-01-27 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: Alcoholism; Delirium; Magnesium Deficiency
MeSH Terms: conditions — Alcoholism; Delirium; Magnesium Deficiency | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Usual care (i.e. without any restriction of drug therapy) plus oral tablet magnesium supplementation: 426.6mg of magnesium per day three times daily (i.e. 142.2 mg for each shot) throughout the study (i.e. fifteen days). In case of diarrhea, nearly half-dosage will be used (i.e. 189.6mg).
  Interventions: Drug: Magnesium
- Control (Placebo Comparator): Usual care (i.e. without any restriction of drug therapy) plus oral placebo, totally similar to the verum, three times daily throughout the study (i.e. fifteen days). In case of diarrhea, nearly half-dosage will be used.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Magnesium — Usual care (i.e. without any restriction of drug therapy) plus oral tablet magnesium supplementation: 426.6mg of magnesium per day three times daily (i.e. 142.2 mg for each shot) throughout the study (i.e. fifteen days). In case of diarrhea, nearly half-dosage will be used (i.e. 189.6mg).
  Arms: Intervention
Drug: Placebo Oral Tablet — Usual care (i.e. without any restriction of drug therapy) plus oral placebo, totally similar to the verum, three times daily throughout the study (i.e. fifteen days). In case of diarrhea, nearly half-dosage will be used.
  Other Names: Placebo
  Arms: Control

SUMMARY:
This study examine the efficacy of oral magnesium supplementation as an adjuvant therapy for decreasing intensity of alcohol withdrawal symptoms among inpatients requiring pharmacological treatment of their AWS. This double blind randomized multicenter clinical trial planned to treat half of participants as usal plus placebo and the other half as usual plus magnesium.

DETAILED DESCRIPTION:
Alcohol withdrawal syndrome (AWS) is a frequent and potentially fatal outcome. It is crucial to treat AWS in order to reduce symptoms severity, to prevent severe complications and to increase patient motivation to maintain long-term alcohol abstinence. Clarify the relevance of oral magnesium supplementation as a routine adjuvant therapy of AWS can give rise to a major evolution of guidelines regarding management of alcohol use disorder and make AWS more comfortable for hundred thousand patients.

Magnesium acts as a competitor of glutamate on NMDA receptor binding site, limiting glutamate toxicity leading to AWS. Previous findings suggested a correlation between AWS intensity and hypomagnesaemia degree, and an increased risk of severe AWS (i.e. delirium tremens and seizure) when there is deep depletion. In addition to magnesium role as a glutamatergic modulator via an NMDA-receptor antagonism activity, magnesium may also modulate GABAergic neurotransmission and affect numerous transduction pathways, including proteinkinase C, possibly influencing the access of corticosteroids to the brain.

Moreover, magnesium has been found to be a cofactor required for thiamine-dependent enzymes whereas thiamine supplementation is crucial to prevent from Wernicke's encephalopathy in the treatment of AWS. Finally, magnesium supplementation could help to reduce benzodiazepines use.

The primary endpoint is the between-group absolute difference of the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) score change from baseline, 3 days after randomization.

The secondary endpoints are:

a Total benzodiazepine consumption compared between experimental and control groups throughout the duration of the study (i.e. 15 days); b Time required to obtain a total score of 0 at the CIWA-Ar compared between experimental and control groups; c Rate of patients experiencing seizures and delirium tremens during the study compared between intervention and control groups; d Stratify results of the Primary endpoint following score at the Charlson Comorbidity Index; e Stratify results of the Primary endpoint by age; f Number of participants who left the hospital against medical advice during the study compared between experimental and control groups; g Number of participants who made an appointment in an addiction unit during the study (i.e. before the last follow-up point, 15 days after baseline), compared between experimental and control groups after stratification following AUD duration and number of previous addiction healthcare; h Patient Satisfaction Questionnaire-18 (PSQ-18) scores at the last follow-up point (i.e. days after baseline) compared between experimental and control groups; i Total plasmatic or serum magnesium concentration changes between baseline, 3 days after baseline, and 7 days after baseline; j Rate of all adverse events occurred during the study incidence compared between experimental and control groups;

Practical procedure:

Patients recruited are inpatients, hospitalized whatever the main reason for hospitalization (i.e. alcohol withdrawal syndrome or other reason). Inclusion visit starts with signature of informed consent, then confirms the eligibility and finally, ends with randomization and administration of the first dose of treatment. Patients are followed 15 days after baseline. Total plasmatic or serum magnesium concentration is dosed at baseline, 3 days and 7 days. In addition to CIWA-Ar and AUDIT, the following assessments are performed at baseline: Charlson comorbidity index, DIGS, SCL-90, MINI. We will use tablets of 465.4 mg of magnesium lactate dehydrate (Magnespasmyl©), which corresponds to 47.4mg of magnesium (i.e. 1.9mmol of magnesium per tablet). These tablets will be prescribed as follows: 3 tablets three times per day. In case of diarrhea, nearly half-dosage will be used until the end of the follow-up (i.e. 189.6mg per day, 3 times a day as follows: 1 tablet, 2 tablets, 1 tablet). Patients will be informed that treatment is to be taken during meals and to avoid sodas during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients, men and women (i.e. age>18 years and <75 years) ;
* Current AWS according to DSM-5 criteria;
* Score at the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) >8;
* Written informed consent to participate in the study;
* Affiliation to the French Social Security Health Care plan.

Exclusion Criteria:

* Age less than 18 or greater than 75;
* Hemodynamic failure;
* Arythmia;
* Lack of fulfilling AWS criteria according to DSM-5;
* Score at the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) <=8;
* Benzodiazepine misuse according to the opinion of the investigator;
* Substance use disorder according to the opinion of the investigator, regarding licit and illicit substances, except for tobacco;
* Pregnancy or breast-feeding;
* Unable to take oral medications;
* Creatinine clearance < 45mL/min less than 6 months old. If there is no dosage in the last 6 months, creatinine clearance must be <30mL/min at inclusion (creatinine clearance computed according to the Cockcroft-Gault Equation);
* Cognitive disorders already known at inclusion that impair the informed consent, including dementia (except for acute withdrawal delirium), according to the opinion of the investigator;
* Psychiatric disorder requiring hospitalization or specific cares in emergency (e.g. suicidal crisis, acute psychotic episode);
* Magnesium supplementation (regardless the type of delivery) within 3 months prior to inclusion;
* Actual quinidine intake;
* No written informed consent to participate in the study;
* Patient under tutorship or curatorship;
* Hypersensitivity to Magnespasmyl® or to any of its excipients (including sucrose) or to lactose (placebo excipient).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Between-group absolute difference of the CIWA-Ar score (revised clinical institute withdrawal assessment for alcohol scale) change from baseline | 3 days after randomization

SECONDARY OUTCOMES:
Total benzodiazepine consumption compared between experimental and control groups throughout the duration of the study | 15 days after randomization
The delay compared between experimental and control groups until having a total score of 0 at the CIWA-Ar | 15 days after randomization
The rate of patients experiencing seizures and delirium tremens during the study compared between intervention and control groups | 15 days after randomization
Between-group absolute difference of the CIWA-Ar score change from baseline, considering two subgroups: score at the Charlson Comorbidity Index (CCI) min-score at the CCI median versus score score at the CCI median-score at the CCI min | 3 days after randomization
Between-group absolute difference of the CIWA-Ar score (revised clinical institute withdrawal assessment for alcohol scale) change from baseline considering two subgroups: 18-59 years versus 60-75 years | 3 days after randomization
The number of participants who left the hospital against medical advice during the study compared between intervention and control groups | 15 days after randomization
The number of participants who made an appointment in an addiction unit during the study compared between intervention and control groups after stratification following alcohol use disorder (AUD) duration and number of previous addiction healthcare | 15 days after randomization
Patient Satisfaction Questionnaire-18 scores at the last follow-up point compared between experimental and control groups | 15 days after randomization
Total plasmatic or serum magnesium concentration changes between baseline,3 days after baseline, and 7 days after baseline, compared between intervention and control groups | 3 days and 7 days after randomization
Rate of all adverse events occurred during the study and compare their incidence between intervention and control groups | 15 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Limosin, M.D., Ph.D., Principal Investigator — Assistance Publique-Hôpitaux de Paris (AP-HP)
Locations (11):
- France (11):
  - Hôpital Emile ROUX, Limeil-Brévannes
  - Hôpital Louis Mourier, AP-HP, Colombes, Île-de-France Region
  - Clinique des Platanes, Épinay-sur-Seine, Île-de-France Region
  - Hôpital Corentin Celton, AP-HP, Issy-les-Moulineaux, Île-de-France Region
  - Institut MGEN de la Verriere, Le Mesnil-Saint-Denis, Île-de-France Region
  - Institut MGEN la Verriere-service SSR addictologie, Le Mesnil-Saint-Denis, Île-de-France Region
  - Clinique des maladies mentales et de l'encéphale, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou-Service de chirugie orthopédique, AP-HP, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou-Service de médecine interne, AP-HP, Paris, Île-de-France Region
  - Hôpital européen Georges-Pompidou-Service hépato-gastroentérologie, Paris, Île-de-France Region
  - Centre Hospitalier des quatre villes, Sèvres, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No